CLINICAL TRIAL: NCT03418428
Title: Surgical Gastric Cancer Treatment: Influence on Intestinal Microbiome
Brief Title: Intestinal Microbiome After Gastrectomy
Acronym: DiGMA
Status: Completed | Type: Observational
Sponsor: Vilnius University (Other)
Collaborators: Medical University of Graz (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rimantas Bausys, Medical Doctor, Vilnius University
Other Study IDs: DiGMA_2018
Record Dates: First submitted 2018-01-02; First posted 2018-02-01 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Test group: Patients who underwent total or subtotal gastrectomy for the treatment of gastric cancer
- Control group 1: Patients who underwent endoscopic mucosal resection/submucosal dissection for the treatment of gastric cancer
- Control group 2: In-house relatives of Test group and Control group 1 participants
- Control group 3: Patients with long-term history of proton pump inhibitor usage

SUMMARY:
The gastric barrier plays a major role in the maintanance of the distal intestinal microbiome composition. It has been shown before that the use of gastric acid suppression medication, such as proton pump inhibitors, are associated with distinctive alterations of the intestinal microbiome. Foremost, the invasion of predominantly oral bacteria, like Veillonella and Streptococcus species, were a resurring finding in previous reports.

Gastric cancer treatment includes the total or subtotal resection of the stomach which can influence the gastric acid production. However, the influence by alterations in gastric milieu after this treatment on the composition of the intestinal microbiome is not well studied.

Therefore, the intestinal microbiome of patients after total or subtotal gastrectomy and its influence on intestinal inflammation and gut permeability will be studied.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and above
* history of radical removal of gastric cancer (Test group and Control group 1) or PPI (Control group 3)
* informed consent

Exclusion Criteria:

* chemotherapy or radiotherapy 12 months prior to inclusion
* gastric stump cancer
* usage of antibiotics, pro- pre or synbiotics, H2-blocker 1 month prior to inclusion
* PPI use (except for Control group 3) 1 month prior to inclusion
* history of radical removal of gastric cancer (Control group 2-3)
* history of gastrointestinal tract resections (other than gastric)
* recurrence of gastric cancer
* current non-gastric malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Test group: Patients with a history of gastric cancer surgery, without the current use of PPI and no recurrence of gastric cancer and a minimum of 12 months since the last adjuvant treatment Control group 1: Patients with a history of endoscopic resection of gastric cancer, without the current use of PPI and no recurrence of gastric cancer Control group2: Healthy volunteers recruited from relatives of study participants (Test group and Control group 1), without the current use of PPI Control group 3: Patients with a history of long-term PPI usage (6 months) without a history of gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Intestinal microbiome composition | 5 years after surgery
  Significant differences in the beta-diversity of the intestinal microbiome between Test group and Control groups

SECONDARY OUTCOMES:
Intestinal microbiome composition (II) | 5 years after surgery
  Significant differences in the alpha-diversity of the intestinal microbiome between Test group and Control groups
Fecal calprotectin | 5 years after surgery
  Significant differences in intestinal inflammation measured by fecal calprotectin between Test group and Control groups
Fecal zonulin | 5 years after surgery
  Significant differences in intestinal permeability measured by fecal zonulin between Test group and Control groups
Serum LPS | 5 years after surgery
  Significant differences in serum LPS between Test group and Control groups
Serum sCD14 | 5 years after surgery
  Significant differences in serum sCD14 between Test group and Control groups
Serum LBP | 5 years after surgery
  Significant differences in serum LBP between Test group and Control groups
Serum sCD163 | 5 years after surgery
  Significant differences in serum sCD163 between Test group and Control groups
Serum sMR | 5 years after surgery
  Significant differences in serum sMR between Test group and Control groups
Serum CRP | 5 years after surgery
  Significant differences in serum CRP between Test group and Control groups
Serum DAO | 5 years after surgery
  Significant differences in serum DAO between Test group and Control groups

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided
The use of sequence data repositories is planed

REFERENCES:
- [Derived] Horvath A, Bausys A, Sabaliauskaite R, Stratilatovas E, Jarmalaite S, Schuetz B, Stiegler P, Bausys R, Stadlbauer V, Strupas K. Distal Gastrectomy with Billroth II Reconstruction is Associated with Oralization of Gut Microbiome and Intestinal Inflammation: A Proof-of-Concept Study. Ann Surg Oncol. 2021 Feb;28(2):1198-1208. doi: 10.1245/s10434-020-08678-1. Epub 2020 Jun 5. PMID 32504369